CLINICAL TRIAL: NCT02991794
Title: Prospective, Multi-centre, Non-interventional Trial on Laparoscopic Radical PROSTatectomies Using EinsteinVISion® 3D Visualization System
Brief Title: Prostatectomies Using Einstein Vision® 3D
Acronym: PROSTEVIS
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1607
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Prostate Carcinoma
Keywords: prostatectomy; laparoscopy; 3D visualization; learning curve; anastomosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EinsteinVision 3D visualization system — Elective laparoscopic radical prostatectomy due to histologically proven prostate cancer using EinsteinVision® 3D visualization system.

SUMMARY:
The aim of the study is collecting clinical data on the learning curve of different surgeons using the EinsteinVision® 3D visualization system in laparoscopic radical prostatectomies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned radical prostatectomy prostatectomy because of histologically proven prostate cancer using EinsteinVision®
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Previous TURP (= transurethral resection of the prostate)
* Previous operations on the sigmoid colon or rectum (e.g. because of carcinoma, perforation, diverticulum)
* BMI > 35 kg/m²
* Participation in another clinical study
* Representation by a legal guardian or under involuntary commitment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Time needed to perform the vesicourethral anastomosis using EinsteinVision® in a group of different surgeons [min. sec.] | Intraoperatively
  learning curve of different surgeons with diverse level of experience using EinsteinVision® 3D visualization system

SECONDARY OUTCOMES:
Intraoperative blood loss [ml] | Intraoperatively
Intraoperative blood transfusions [quantity] | Intraoperatively
Postoperative blood transfusions [quantity] | Postoperatively
Intraoperative incidence of complications [percentage] | Intraoperatively
  (e.g. bleedings, Trauma of ureter)
Postoperative incidence of complications [percentage] | During stay in Hospital (5-12 days postoperatively)
  (e.g. Ileus, venous thrombo-embolic events, wound infection, bleedings)
Surgeon's experience with different operation methods and application systems | After first intervention for each hospital and after study completion, an average of 1 year later
  using a questionnaire at the beginning (First Patient In) and the end of the study (Last Patient In)
Patient's quality of life | Preoperatively, 5-12 days postoperatively, 3 months, 6 months, 12 months postoperatively
  Pre- and postoperative patient's quality of life using the questionnaire EQ-5D-5L
  The following dimensions are assessed:
  * Mobility
  * Self-care
  * Usual activities
  * Pain / discomfort
  * Anxiety / depression
  * Health
Operation time [min.] | Intraoperatively
Intraoperative usability of the device | Intraoperatively
  using a questionnaire containing different dimensions and a 5-point assessment level (Likert Scale: 1 = excellent, 5 = unacceptable).
  The following dimensions are assessed:
  * Control
  * Expenditure of energy
  * Image quality
  * Overall satisfaction
Incontinence after catheterization [percentage] | During stay in Hospital (5-12 days postoperatively)
Postoperative hospital stay [days] | During stay in Hospital (5-12 days postoperatively)
Return to erectile function [percentage] | 12 months
Return to continence function [percentage] | 12 months
Incontinence pads/pants per day [quantity] | 5-12 days postoperatively, 3 months, 6 months, 12 months postoperatively
Postoperative patient satisfaction | 5-12 days postoperatively, 3 months, 6 months, 12 months postoperatively
  using a 10-point assessment level (1 = completely dissatisfied, 10 = completely satisfied)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Sana Klinikum Offenbach, Offenbach
  - medius Klinik Ostfildern-Ruit, Ostfildern

IPD SHARING:
Plan to Share IPD: No